CLINICAL TRIAL: NCT02151266
Title: The Feasibility of Exercise and Cognitive Retraining to Improve Memory, Attention and Concentration in Heart Failure.
Brief Title: Exercise and Cognitive Retraining to Improve Cognition in Heart Failure.
Acronym: EXCITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rebecca Gary, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00060752; P30NR014134 (NIH)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
Keywords: Heart failure; Exercise; Cognitive training
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Exercise; Walking; Pliability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exercise and Cognitive retraining (Experimental): Aerobic exercise; Computerized cognitive retraining program; Heart failure education; Home visits; telephone follow-up.
  Interventions: Behavioral: Exercise and Cognitive retraining
- Exercise only (Experimental): Each participant will be provided with an individualized target heart rate (THR)zone based on treadmill results. Under the supervision of a research nurse, participants will begin the walking sessions at 60% of THR and increase to 70% by week 5. Participants will walk a minimum of 5 times per week for a duration of 30 minutes.
  Interventions: Behavioral: Exercise Only
- Stretching and Flexibility (Sham Comparator): Stretching and flexibility movements; heart failure education; home visits; telephone follow-up.
  Interventions: Behavioral: Stretching and Flexibility

INTERVENTIONS:
Behavioral: Exercise and Cognitive retraining — Walking 5 times per week at moderate intensity; cognitive retraining one-hour 2 times per week.
  Other Names: Aerobic exercise; walking and computerized cognitive retraining program
  Arms: Exercise and Cognitive retraining
Behavioral: Exercise Only
  Arms: Exercise only
Behavioral: Stretching and Flexibility
  Arms: Stretching and Flexibility

SUMMARY:
Cognitive impairment (CI) is a prevalent problem in persons with HF heart failure (HF) and is associated with adverse clinical outcomes, higher mortality and poorer quality of life. Studies designed to attenuate or alleviate CI in persons with HF are limited, and evidenced based guidelines for screening and provision of care are practically nonexistent. Improvement in cognition has been reported following some therapies in HF and is thought to be the consequence of enhanced cerebral perfusion and oxygenation, suggesting that CI may be amenable to intervention in this population. Exercise is documented to increase cerebral perfusion and oxygenation by promoting neuroplasticity and neurogenesis, and, in turn, cognitive functioning. Brain derived neurotrophic factor (BDNF) is a key mechanism underlying the effect of exercise, but most studies of BDNF have not included individuals with CI or chronic illness populations, and its relationship to cognitive outcomes in HF is unknown. Cognitive retraining techniques, originally developed to treat traumatic brain injury, have also shown efficacy in broader neurologically-affected conditions and may provide added benefit to that of exercise. Animal studies suggest exercise and plasticity-based cognitive training could act synergistically through different neural mechanisms to have a more pronounced and positive impact on cognitive outcomes than either approach alone; but this has not been previously tested as an intervention to improve CI. The proposed feasibility study is designed to test the acceptability and limited efficacy of a combined exercise (Ex) and cognitive training (CT) program to improve CI in stable NYHA class II and III HF patients compared to either exercise alone or a no-intervention, attention-control group. Findings will be used to support the development of a future, large scale study to test the efficacy of this intervention to improve cognitive functioning, quality of life, and physiological markers of improved brain function in HF. In addition, we have an optional sub-study that participants may participate in order to further our understanding of biomarkers of inflammation and gen e expression before and after exercise.

DETAILED DESCRIPTION:
Persons with heart failure (HF) have a four-fold greater likelihood of developing cognitive impairment (CI) than their age matched healthy counterparts, placing them at high risk for adverse clinical outcomes, poorer quality of life (QOL) and higher mortality. CI is a subtle but measurable deficit in one or multiple cognitive domains; it is a deficit greater than cognitive losses associated with normal aging. The few studies that have documented CI in HF are inconsistent. Few have used standard neuropsychological testing, and little is known about change in cognitive function over time in HF. Further, if CI is detected, there are currently no effective or evidenced-based guidelines to help restore or improve cognition in this population.Despite the aging population and projected rise of CI in HF, only 2 small intervention studies have been documented, indicating a critical need for further research in this area.

The etiology of CI in HF is not fully understood, but several underlying mechanisms are consistently reported: reduced cerebral perfusion and oxygenation, brain structural changes (i.e., hippocampal damage, atrophy, loss of gray matter), and micro emboli.Clinical studies have shown that CI is improved after cardiac transplantation and is modifiable with standard therapies that improve cardiac output, oxygenation, fluid overload, and systemic and cerebral perfusion; these findings are inconsistent and anecdotal. The ability to positively influence cognitive function has important implications for patient adherence to a complex self-care regimen and the development of interventions that may partially reverse CI.

Exercise improves clinical outcomes in HF by altering the deleterious peripheral and central mechanisms that contribute to HF exacerbations, worsen symptom severity, and lead to poor clinical outcomes. Less is known about the effect of exercise on cognitive function. Animal research has provided the most compelling evidence that exercise positively affects neuronal growth and the neural systems involved in learning and memory. Similar human findings have emerged; recent advances in neuroimaging support that participation in regular exercise leads to specific changes in brain structure and function. Exercise is also thought to enhance brain plasticity. BDNF appears to play a crucial role in this process: when BDNF levels increase following exercise, cognitive function improves. The association between exercise, BDNF and cognitive function has not been previously reported in HF. This feasibility study will clarify these important relationships and increase the potential for improving clinical outcomes in a future trial.

Neurogenesis and neuroplasticity are means for the brain to recover from poor perfusion and oxygen deprivation such as that occurring in HF. Animal studies again provide the strongest evidence to date for using cognitive training (CT) to promote better cognitive functioning and provide a rationale for why a combined exercise and CT approach may be superior to monotherapy. Animal studies show that, like exercise, learning tasks and performing cognitively stimulating activities also increase BDNF levels and improve learning and memory. The effect of BDNF on brain function due to exercise however, is thought to be different from that occurring with CT. Exercise increases the proliferation and division of neuronal cells through BDNF, whereas CT appears to promote cell survival,suggesting a synergistic relationship may exist with greater benefit obtained when both are used together. The combination of exercise and plasticity-based CT has not been previously tested in HF or in other populations as an intervention for improving cognitive outcomes, but may be most optimal for targeting the underlying mechanisms for CI in HF. The proposed feasibility study is designed to test the acceptability, implementation and limited efficacy of a combined exercise (Ex) and cognitive training (CT) intervention in stable NYHA class II and III heart failure patients with cognitive impairment. A total of 60 participants will be randomized to one of three study arms: Ex/CT (N=20), Ex-alone (N=20), and attention control (N=20). The study aims are:

Aim 1: To evaluate the feasibility of a 3-arm intervention (ExCT, Ex, AC) in heart failure patients with CI.

Aim 1a. To test the acceptability and implementation of each study arm. Aim 2: To ascertain limited efficacy of the 3-arm intervention on changes in cognitive abilities Aim 3: To ascertain limited efficacy of the 3-arm intervention to improve cerebral oxygenation, physiological status, physical function and QOL.

ELIGIBILITY:
Inclusion Criteria:

men and women between the ages of 40 and 75; English speaking; live independently within a 60 mile radius of Atlanta; meet education corrected cut-offs on the MMSE indicating cognitive impairment (score of 20 for 8-9 yrs of schooling; 22 for 10-12 yrs of schooling; 23 for >12 yrs) have a computer with internet connection; documented medical diagnosis of NYHA class II or III systolic. Left ventricular ejection fraction (LVEF) ≥ 10% that is documented within the last year by echocardiogram, cardiac catheterization ventriculography or radionuclide ventriculography; Receiving medication therapy for HF according to American College of Cardiology (ACC) American Heart recommendation guidelines for at least 8 weeks prior to study enrollment.

-

Exclusion Criteria:

NYHA class I or IV; change in HF therapy within 8 weeks; worsening HF symptoms within last 5 days; unstable angina; renal insufficiency (serum creatinine > 3.o mg/dL); fixed rate pacemaker; uncontrolled hypertension; not involved in any structured exercise program or exercising 3 or more times per week for a minimum of 30 minutes and; not hospitalized within the last 30-days; not diagnosed with any neurological disorder that may interfere with cognitive function; Beck Depression Inventory II (BDI-II) score greater than 25; any disorder interfering with exercise participation.

-

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-07; Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University Heart Failure Clinics, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Gary RA, Paul S, Corwin E, Butts B, Miller AH, Hepburn K, Waldrop D. Exercise and Cognitive Training Intervention Improves Self-Care, Quality of Life and Functional Capacity in Persons With Heart Failure. J Appl Gerontol. 2022 Feb;41(2):486-495. doi: 10.1177/0733464820964338. Epub 2020 Oct 13. PMID 33047625
- [Derived] Gary RA, Paul S, Corwin E, Butts B, Miller AH, Hepburn K, Williams B, Waldrop-Valverde D. Exercise and Cognitive Training as a Strategy to Improve Neurocognitive Outcomes in Heart Failure: A Pilot Study. Am J Geriatr Psychiatry. 2019 Aug;27(8):809-819. doi: 10.1016/j.jagp.2019.01.211. Epub 2019 Feb 1. PMID 30910420

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Only: Each participant will be provided with an individualized target heart rate (THR)zone based on treadmill results. Under the supervision of a research nurse, participants will begin the walking sessions at 60% of THR and increase to 70% by week 5. Participants will walk a minimum of 5 times per week for a duration of 30 minutes.
  Exercise Only
- Stretching and Flexibility: Stretching and flexibility movements; heart failure education; home visits; telephone follow-up.
  Stretching and Flexibility
Period: Overall Study
Arm/Group | Exercise and Cognitive Retraining | Exercise Only | Stretching and Flexibility
Started | 19 | 29 | 21
Completed | 11 | 14 | 14
Not Completed | 8 | 15 | 7
Not completed — Lost to Follow-up | 1 | 4 | 1
Not completed — Did NOT receive intervention | 3 | 6 | 2
Not completed — Not able to exercise | 4 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise and Cognitive Retraining | Exercise Only | Stretching and Flexibility | Total
Number analyzed (Participants) | 19 | 29 | 21 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (11) | 60 (10) | 63 (9) | 61 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 8 | 37
  Male | 7 | 12 | 13 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 16 | 9 | 38
  White | 4 | 12 | 11 | 27
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 29 | 21 | 69

OUTCOME MEASURES:

1. Primary Outcome: Verbal Memory Score Change
Description: List Learning (0-40), List Recall (0-10), and List Recognition (0-20) sections from the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) are used to assess Verbal memory.The range of scores for each section are in parentheses. Higher scores reflect better verbal memory. Scores are averaged for a total Verbal memory score, then converted to Z-score.
  Z-scores are used when neurocognitive test scores use different measurement scales, e.g., time to completion and number correct. This allows to report performance in a straightforward manner, with low and high scores reflecting poor and good performance consistently across different types of tests, and to provide interpretation of a person's performance in comparison to a group. For interpretive purposes, a z-score has a mean of 0 and a standard deviation of 1. This means that an individual who has a z-score of 1.5 is performing one and a half standard deviations above the group to which he/she is compared.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise and Cognitive Retraining | Exercise Only | Stretching and Flexibility
Number analyzed (Participants) | 11 | 14 | 14
score on a scale
  baseline | -0.08 (0.20) | -0.08 (0.15) | 0.18 (0.19)
  3 months | -0.47 (0.21) | 0.14 (0.18) | 0.37 (0.20)
  6 months | -0.20 (0.21) | 0.07 (0.19) | 0.25 (0.22)

2. Secondary Outcome: Functional Capacity
Description: Functional capacity will be assessed by six-minute walk across all 3 arms of the study.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Exercise and Cognitive Retraining | Exercise Only | Stretching and Flexibility
Number analyzed (Participants) | 11 | 14 | 14
meters
  baseline | 324.1 (19.2) | 355.1 (15.9) | 337.6 (18.5)
  3 months | 311.1 (20.0) | 358.8 (16.9) | 388.4 (20.2)
  6 months | 321.2 (20.2) | 374.9 (18.7) | 374.9 (20.6)

3. Other Pre Specified Outcome: Peak V02
Description: To evaluate change in cardio-respiratory fitness Peak V02 was assessed at baseline and 3 months using a motorized treadmill test across 3 arms of the study
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Exercise and Cognitive Retraining | Exercise Only | Stretching and Flexibility
Number analyzed (Participants) | 11 | 14 | 14
mL/kg/min
  3 months | 15.9 (1.3) | 16.2 (1.0) | 19.3 (1.2)
  baseline | 15.3 (1.3) | 16.0 (1.0) | 19.3 (1.1)

4. Primary Outcome: Visual Memory Score Change
Description: Visual memory will be assessed using Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). RBANS figure recall requires the participant to remember a recent figure and redraw it from memory. The range of possible scores is 0-20. Scores are averaged, and then converted to z score.
  Z-scores are used when neurocognitive test scores use different measurement scales, e.g., time to completion and number correct. This allows to report performance in a straightforward manner, with low and high scores reflecting poor and good performance consistently across different types of tests, and to provide interpretation of a person's performance in comparison to a group. For interpretive purposes, a z-score has a mean of 0 and a standard deviation of 1. This means that an individual who has a z-score of 1.5 is performing one and a half standard deviations above the group to which he/she is compared.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: z scores
Arm/Group | Exercise and Cognitive Retraining | Exercise Only | Stretching and Flexibility
Number analyzed (Participants) | 11 | 14 | 14
z scores
  baseline | -0.09 (0.23) | -0.17 (0.18) | 0.29 (0.22)
  3 months | -0.21 (0.24) | 0.08 (0.21) | 0.18 (0.24)
  6 months | -0.90 (0.25) | -0.14 (0.23) | 0.32 (0.25)

5. Primary Outcome: Change in Processing Speed/Attention Score
Description: RBANS coding (0-89) Color Trails 1 (timed test, 1-5 minutes) measures attention. The length of time to complete each part is recorded; lower raw scores reflect better processing speed and attention. Lower raw scores reflect better processing speed and attention. Scores are averaged for a total score, then converted to Z scores.
  Z-scores are used when neurocognitive test scores use different measurement scales, e.g., time to completion and number correct. This allows to report performance in a straightforward manner, with low and high scores reflecting poor and good performance consistently across different types of tests, and to provide interpretation of a person's performance in comparison to a group. For interpretive purposes, a z-score has a mean of 0 and a standard deviation of 1. This means that an individual who has a z-score of 1.5 is performing one and a half standard deviations above the group to which he/she is compared.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: z scores
Arm/Group | Exercise and Cognitive Retraining | Exercise Only | Stretching and Flexibility
Number analyzed (Participants) | 11 | 14 | 14
z scores
  baseline | -0.09 (0.11) | -0.02 (0.10) | 0.12 (0.11)
  3 months | -0.09 (0.12) | 0.13 (0.11) | -0.01 (0.13)
  6 months | 0.20 (0.13) | -0.02 (0.12) | -0.18 (0.14)

6. Primary Outcome: Change in Working Memory Score
Description: Digit Span Forward (0-16), Digit Span Backwards (0-16), Digit Span Sequencing (0-16) and Letter Number Sequencing (0-48) sections from the Wechsler Adult Intelligence Scale - Fourth Edition are used to assess Working Memory. The range of possible scores for each section are in parentheses. The Digit Span subtest require the repetition of verbally presented series of numbers that increase in length; trials include the repeating of numbers in forward, backward, and numerical order. The Letter-Number sequencing test requires the repeating strings of letters and numbers in numerical and then in alphabetical order. Color Trails Test (CTT) Part 2, participants rapidly connect numbered circles in sequence while alternating between pink and yellow circles. Higher scores reflect better outcome. Scores reflect number correct and are averaged for total correct Working Memory score; are then converted to Z-score.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: z scores
Arm/Group | Exercise and Cognitive Retraining | Exercise Only | Stretching and Flexibility
Number analyzed (Participants) | 11 | 14 | 14
z scores
  baseline | -0.04 (0.12) | 0.09 (0.10) | -0.07 (0.12)
  3 months | -0.03 (0.13) | 0.12 (0.11) | -0.16 (0.13)
  6 months | -0.15 (0.13) | 0.10 (0.12) | -0.03 (0.14)

7. Primary Outcome: Change in Reaction Time
Description: Scores are automatically calculated via the scoring software embedded within the CalCap and are standardized based on age and education level norms. Normative data are stratified by both age (20-34, 35-44, 45+) and education (< 16 years, 16 years, > 16 years). Lower scores reflect slower reaction time and higher scores reflect faster reaction time. Scores are automatically converted to age/education based standard scores and are reported as a T-score.
  T-scores (as Z-scores) are used when neurocognitive test scores use different measurement scales, e.g., time to completion and number correct. This allows to report performance in a straightforward manner, with low and high scores reflecting poor and good performance consistently across different types of tests, and to provide interpretation of a person's performance in comparison to a group.
Time Frame: Baseline, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: t scores
Arm/Group | Exercise and Cognitive Retraining | Exercise Only | Stretching and Flexibility
Number analyzed (Participants) | 11 | 14 | 14
t scores
  baseline | 0.14 (0.22) | 0.11 (0.18) | 0.29 (0.22)
  3 months | -0.05 (0.25) | 0.07 (0.21) | 0.18 (0.24)
  6 months | 0.02 (0.24) | -0.13 (0.23) | 0.30 (0.26)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Exercise and Cognitive Retraining | Exercise Only | Stretching and Flexibility
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/29 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/29 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/29 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT02151266/Prot_SAP_000.pdf